CLINICAL TRIAL: NCT03905200
Title: Study on the Value of Three-dimensional Speckle Tracking Technique in the Diagnosis and Follow-up of Coronary Heart Disease
Brief Title: Study on the Value of Three-dimensional Speckle Tracking Technique
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Fang Wang, Professor, Beijing Hospital
Other Study IDs: Z161100000516053
Record Dates: First submitted 2019-03-31; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Echocardiography, Three-Dimensional; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- coronary artery disease: Patients who were diagnosed with coronary heart disease at admission and planned to undergo coronary angiography
  Interventions: Diagnostic Test: 3D-speckle tracking imaging

INTERVENTIONS:
Diagnostic Test: 3D-speckle tracking imaging — The strain peak value and strain peaking time of each segment (including 16 segments) of the left ventricular myocardium can be obtained by 3d-sti technology.

SUMMARY:
For a long time, it has been hoped that doctors could screen and diagnosis of coronary heart disease through non-invasive imaging techniques, so as to maximize the benefit/risk ratio of patients. This trial is to explore the screening and diagnostic value of three-dimensional speckle tracking technology for coronary heart disease, and the evaluation value of 3D speckle track image(3D-STI) technology for cardiac function improvement after coronary intervention, and to seek reliable, accurate and quantifiable non-invasive imaging examination for the diagnosis, follow-up and prognosis of coronary heart disease.

In this study, coronary angiography is taken as the "gold standard", and 3d-STI echocardiography technology is proposed to combine with clinical characteristics of subjects for joint diagnosis, so as to evaluate the value of 3d-sti technology in the diagnosis of coronary heart disease.

Patients were followed up with echocardiography after interventional treatment to explore the feasibility of 3D-STI technology in evaluating cardiac function improvement.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with coronary heart disease
* patients underwent coronary angiography with or without PCI

Exclusion Criteria:

* patients with non-sinus rhythm
* patients with severe heart valvular disease
* patients with severe cardiomyopathy
* patients with congenital heart disease
* patients with severe heart failure stage
* patients with acute myocardial infarction occurred during follow-up
* patients with other extremely severe illness
* patients whose images are not clear enough to mark the endocardium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to reference, the area under the ROC curve of 3d-STI strain peak and strain peaking time for the diagnosis of coronary heart disease is about 0.65.In this study, it is expected that the combined diagnosis model can increase the area under the ROC curve to the level of 0.85, and the standard deviation of the area under the ROC curve is estimated to be 0.5. In order to get 85% assurance, we plan to include 827 subjects.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular myocardial viability | half an hour
  By measuring the strain and time to peak, the left ventricular myocardial viability was finally evaluated. Left ventricular local ventricular viable myocardium was quantitatively analyzed in patients .Aimed to detect the myocardial ischaemia and viability. The data of strain and time to peak were measured using the three-dimensional speckle tracking model.
  In apical four-chamber view, make sure the endocardium, mitral valve ring and apex imaging is clear, mark the left and right mitral valve ring and apex spot . After automatic ultrasonic echo spot tracked, software can delineate endocardial curve, and automaticaly calculate the left ventricular myocardial segments strain and time to peak.
  The strain peaks of each segment (including 16 segments) of the myocardium of the left ventricle included four strain peaks: RS, CS, LS and AS

SECONDARY OUTCOMES:
The value of 3D-STI technology on the improvement of left ventricular myocardial function | half a year
  During the 6-month follow-up, 3D-STI technique was used to evaluate the improvement of left ventricular myocardial function compared with conventional parameters like LVEF and NYHA. 3D-STI parameters are the same : strain and peak time .

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Guo Y, Song X, Xu T, Guo H, Yang C, Zhong Y, Li H, Gong J, Wang F. Utilizing machine learning in echocardiographic analysis to distinguish obstructive and non-obstructive coronary artery disease. Int J Cardiol. 2026 Mar 15;447:134121. doi: 10.1016/j.ijcard.2025.134121. Epub 2025 Dec 25. PMID 41455557
- [Derived] Guo Y, Cai YH, Xu T, Song XY, Guo HX, Dong M, Ni D, Li H, Wang F, Xue WF. Echocardiographic video-driven multi-task learning model for coronary artery disease diagnosis and severity grading. Front Bioeng Biotechnol. 2025 Jul 25;13:1556748. doi: 10.3389/fbioe.2025.1556748. eCollection 2025. PMID 40787200
- [Derived] Guo Y, Xia C, Zhong Y, Wei Y, Zhu H, Ma J, Li G, Meng X, Yang C, Wang X, Wang F. Machine learning-enhanced echocardiography for screening coronary artery disease. Biomed Eng Online. 2023 May 11;22(1):44. doi: 10.1186/s12938-023-01106-x. PMID 37170232
- [Derived] Guo Y, Wang X, Yang CG, Meng XY, Li Y, Xia CX, Xu T, Weng SX, Zhong Y, Zhang RS, Wang F. Noninvasive assessment of myocardial work during left ventricular isovolumic relaxation in patients with diastolic dysfunction. BMC Cardiovasc Disord. 2023 Mar 10;23(1):129. doi: 10.1186/s12872-023-03156-4. PMID 36899310